CLINICAL TRIAL: NCT05767294
Title: Epidemiological and Clinical Characteristics of Hospitalized Patients Under 5 Years Old With RSV Infection in Central China, Wuhan
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Sainan Shu, Tongji Hospital, Tongji Medical college, Huazhong University of Science & Technology, Tongji Hospital
Other Study IDs: MISP-100898
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Neonatal
  Interventions: Other: Observation
- 1-3 months old
  Interventions: Other: Observation
- 3-6 months old
  Interventions: Other: Observation
- 6 months-1 year old
  Interventions: Other: Observation
- 1-2 years old
  Interventions: Other: Observation
- 2-5 years old
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — clinical manifestation (body temperature, fever days before admission, cough, red throat/sore throat, runny nose, shortness of breath, wheezing, vomiting), physical signs (auscultation of lungs, X-ray results), length of stay, therapeutic measures (oxygen therapy, ICU admission, antibiotic therapy, etc.)

SUMMARY:
The study will be a multicenter, hospital-based retrospective study. We plan to collect the clinical and laboratory data among all hospitalized ARTI cases in three hospitals in Wuhan from June 1, 2020 to May 31, 2023 and then analyze the epidemiological and clinical characteristics of RSV infection, clarify the gene types of epidemics under 5 years old children after the outbreak in Wuhan, China.

ELIGIBILITY:
Inclusion Criteria:

①Admission age <5 years old

②Clinical diagnosis of acute respiratory tract infections

Exclusion Criteria:

Hospital acquired ARTI

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all hospitalized ARTI cases in three hospitals in Wuhan from June 1, 2020 to May 31, 2023 and then analyze the epidemiological and clinical characteristics of RSV infection, clarify the gene types of epidemics under 5 years old children after the outbreak in Wuhan, China
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with fever | at admission
  number of patients with fever
number of patients with cough | at admission
  number of patients with cough
number of patients with shortness of breath | at admission
  number of patients with shortness of breath
number of patients with shortness of wheeze | at admission
  number of patients with shortness of wheeze
number of patients with shortness of vomit | at admission
  number of patients with shortness of vomit
number of patients with shortness of rale | at admission
  number of patients with shortness of rale
number of patients with shortness of stridor | at admission
  number of patients with shortness of stridor
age | at admission
  age
gender | at admission
  female/male
number of patients with underlying disease | at admission
  underlying disease include immune deficiency, CHD, BPD, BO, bronchiectasis and asthma and so on
Imaging examination results | through study completion, an average of 1 year
  X-Ray/CT
length of hospital stay length of stay length of stay | through study completion, an average of 1 year
  length of hospital stay
number of patients with treatment of antibiotic | through study completion, an average of 1 year
  number of patients with treatment of antibiotic
number of patients with treatment of immunoglobulin | through study completion, an average of 1 year
  number of patients with treatment of immunoglobulin
number of patients with treatment of glucocorticoids | through study completion, an average of 1 year
  number of patients with treatment of glucocorticoids
number of patients with treatment of oxygen inhalation | through study completion, an average of 1 year
  number of patients with treatment of oxygen inhalation
number of patients with treatment of ventilation | through study completion, an average of 1 year
  number of patients with treatment of ventilation
direct medical cost | through study completion, an average of 1 year
  direct medical cost
proportion of different virus genotype | through study completion, an average of 1 year
  virus genotype include A, B and C
F protein gene sequence | through study completion, an average of 1 year
  F protein gene sequence
number of patients infected with bacteria | through study completion, an average of 1 year
  number of patients infected with bacteria
number of patients infected with virus | through study completion, an average of 1 year
  number of patients infected with virus
number of patients infected with fungus | through study completion, an average of 1 year
  number of patients infected with fungus

CONTACTS AND LOCATIONS:
Locations (1):
- department of pediatrics, Tongji hospital, Tongji medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided